CLINICAL TRIAL: NCT03708900
Title: A Phase II, Multicenter, Open-label, Non-comparative Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Tolerability of Osilodrostat in Children and Adolescent Patients With Cushing's Syndrome
Brief Title: Pharmacokinetic (PK), Pharmacodynamic (PD) and Tolerability of Osilodrostat in Pediatric Patients With Cushing's Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCI699C2203; 2018-001522-25 (EudraCT Number)
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cushing Syndrome
Keywords: Cushing's syndrome (CS); LCI699; osilodrostat; Pituitary Gland; Adrenocorticotropic Hormone (ACTH); Urinary Free Cortisol (UFC); mean Urinary Free Cortisol (mUFC)
MeSH Terms: conditions — Cushing Syndrome; Pituitary Diseases | interventions — Osilodrostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LCI699 (osilodrostat) (Experimental): Subjects with cushing's syndrome taking LCI699 (osilodrostat)
  Interventions: Drug: LCI699

INTERVENTIONS:
Drug: LCI699 — osilodrostat (LCI699) is in the form of tablets 1 milligram (mg), 5 mg, and 10mg or in form of capsules 0.1 mg, 0.2 mg, 0.5 mg, 1 mg or 5 mg, both the formulations for oral administration
  Other Names: osilodrostat

SUMMARY:
Multicenter, open-label, non-comparative study to evaluate the pharmacokinetics, pharmacodynamics, and tolerability of osilodrostat in children and adolescent patients with Cushing's syndrome.

DETAILED DESCRIPTION:
The period 1 study duration will be 12 weeks. The study will include a screening period of up to 4 weeks prior to Day 0 (baseline) (to allow for an adequate washout period from any medications that may modify cortisol levels). All subjects being treated with osilodrostat at 12 weeks and obtaining benefit from therapy, per investigator judgment, will be offered participation in an optional 9-month extension period, during which assessment of the PD activity and safety/tolerability of osilodrostat will be done. Patients who do not enter the optional extension period will have a safety follow up visit 4 weeks later.

ELIGIBILITY:
Inclusion criteria

1. Male and female children and adolescents from 2 to < 18 years of age with Cushing's syndrome of endogenous origin: Who have failed surgery (or) who are awaiting surgery (or) for whom surgery is not an immediate option. For patients who are awaiting surgery, the study treatment could be less than 12 weeks.
2. Patients must weigh > 10 kg.
3. The diagnosis of Cushing's syndrome must be confirmed by each of the following:

3a) The clinical criterion of decreasing growth percentiles with increasing weight (as evidenced by the presence of a contrast in height and BMI SD scores, for example a SDS < 0 and BMI SDS > 0, or a strong clinical suspicion of Cushing's syndrome, such as photographic evidence of a change in facial appearance); 3b) Abnormal low-dose (0.5 mg Q6h x 48 hours, or overnight 15mcg/kg [max 1 mg]) dexamethasone suppression test, defined as plasma cortisol levels > 1.8 mcg/dl, at time point 48 hours (0.5 mg Q6h x 48 hours) or 9 to 12 hours (overnight 15mcg/kg [max 1 mg]) after the first dose of dexamethasone; (OR) Midnight serum cortisol levels > ULN, assessed while the patient is sleeping and after pre-cannulation (OR) two samples of late-night salivary cortisol greater than ULN for the assay. 3c)Two 24-hour urinary free cortisol values > 1.3 x ULN;

4. Able to swallow study drug tablets (not crushed or split) or the content of the capsules mixed with water.

5. Parents or legal guardians able to provide consent/assent.

Exclusion Criteria

1. Patients with macroadenoma complicated by compressive symptoms (requiring urgent surgical intervention) or at high risk for compressive symptoms due to mass effect of tumor (concern of corticotroph tumor progression).
2. Insufficient washout period from any other medication used to lower cortisol levels (5 half-lives of any drug).
3. Use of other investigational drugs at the time of enrollment, or within 30 days, or prior to completion of a wash-out duration that is at least 5 half- lives of the drug, at the time of enrollment, whichever is longer. Local regulations may require a longer wash-out period or specify other limitations for participation in an investigational trial, in which case they will be applicable as well.
4. History of hypersensitivity to drugs of the same or similar chemical classes as osilodrostat.
5. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
6. Patients with moderate to severe renal impairment (estimated GFR < 60 mL/min by the Creatinine-based "Bedside Schwartz" equation).
7. Patients with serum ALT and/or AST > 3 x ULN, or total bilirubin > 1.5 x ULN.
8. History of thrombosis.
9. Patients with risk factors for QTc prolongation or Torsade de Pointes, including: 9a) patients with a baseline QTcF > 450 ms 9b) personal or family history of long QT syndrome 9c) concomitant medications known to prolong the QT interval 9d) patients with hypokalemia, hypocalcaemia, or hypomagnesaemia, if not corrected before pre-dose Day 0. In case of uncorrected hypokalemia (<3.5 mEq/L), the screening period may be used to correct hypokalemia prior to starting study drug. Use of potassium supplements and/or mineralocorticoid antagonists is permitted during the study. 9e) Patients with a history of significant cardiovascular disease (based on the opinion of the investigator) such as: structural cardiovascular abnormalities, arrhythmia,
10. Hypertensive patients with uncontrolled blood pressure defined as SBP > 150 and/or DBP > 100 or not optimally treated for hypertension as judged by the investigator.
11. Patients who have undergone any major surgery within 1 month.
12. Patients who have undergone trans-sphenoidal pituitary surgery within 6 weeks prior to screening are not eligible, unless they have clear evidence of persistent hypercortisolism or persistent biochemical changes consistent with Cushing's syndrome.
13. Use of or anticipated use of systemic glucocorticoid medications 1 month prior to screening.
14. Uncontrolled hypothyroidism as evidenced by Free T4 < 0.8 ng/dl.
15. Uncontrolled hyper thyroidism.
16. Diabetic patients with poorly controlled diabetes as evidenced by HbA1c > 8.5 % or not optimally treated for diabetes mellitus as judged by the investigator.
17. Positive pregnancy test in females of childbearing potential.
18. Female patients of childbearing potential who do not agree to use highly effective birth control methods .
19. Pregnant or nursing (lactating) women.
20. Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures. Any severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for the study.
21. Use of concomitant prohibited medications

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2027-07-21 (Estimated); Study Completion 2027-07-21 (Estimated)

PRIMARY OUTCOMES:
Core Study: Evaluate the pharmacokinetics (PK) of osilodrostat using Pharmacokinetic parameters of osilodrostat up to Week 12 in children and adolescents 2 to less than 18 years of age with Cushing's Syndrome | up to Week 12
  evaluate the pharmacokinetics (PK) of osilodrostat in children and adolescents of 2 to less than 18 years of age with Cushing's Syndrome

SECONDARY OUTCOMES:
Core Study: Percentage of patients with normal mean urinary free cortisol (mUFC) at week 3, 6, 9 and week 12 (or end of treatment) | week 3, 6, 9 and week 12 (or end of treatment)
  The assessment in the core period will be done by taking the percentage of patients with normal mUFC at week 6 and week 12 (or end of treatment).
Core Study: Change from baseline in mean urinary free cortisol (mUFC) during the core study period | week 3, 6, 9 and week 12 (or end of treatment)
  The assessment will be done by comparison of change from the baseline in mUFC during core study period on patients
Extension: Efficacy of osilodrostat as measured by mUFC levels up to Month 12 | up to month 12
  The assessment of efficacy of osilodrostat to be measured by change in baseline of mUFC levels up to 12 months on patients
Extension: Efficacy of osilodrostat as measured by mUFC levels up to Month 12 | up to month 12
  The assessment of efficacy of osilodrostat to be measured byproportion of patients with normal mUFC levels at each visit up to 12 months
assessment of the pharmacodynamics, safety and tolerability of osilodrostat. | week 3, 6, 9 and week 12 (or end of treatment)
  Change from baseline in weight in core period
assessment of the pharmacodynamics, safety and tolerability of osilodrostat up to 12 months | up to 12 months
  Change from baseline in weight at each visit in extension period
assessment of the pharmacodynamics, safety and tolerability of osilodrostat.assessment of the pharmacodynamics, safety and tolerability of osilodrostat. | week 3, 6, 9 and week 12 (or end of treatment)
  Change from baseline in body mass index in core period
assessment of the pharmacodynamics, safety and tolerability of osilodrostat.assessment of the pharmacodynamics, safety and tolerability of osilodrostat. | up to 12 months
  Change from baseline in body mass index at each visit in extension period
assessment of the pharmacodynamics, safety and tolerability of osilodrostat. | week 3, 6, 9 and week 12 (or end of treatment)
  Change from baseline in height in core period
assessment of the pharmacodynamics, safety and tolerability of osilodrostat. | up to 12 months
  Change from baseline in height at each visit in extension period

CONTACTS AND LOCATIONS:
Overall Officials: Recordati AG, Study Director — Recordati AG
Locations (15):
- United States (5):
  - University of California San Francisco UCSF, San Francisco, California
  - ABMED Clinical Research Corp, Cape Coral, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - National Institute of Child Health and Human Development, Bethesda, Maryland
  - Texas Valley Clinical Research, Weslaco, Texas
- UZ Brussel, Jette, Brussels Capital, Belgium
- Multiprofile Hospital for Active Treatment Sveta Marina EAD, Varna, Bulgaria
- France (3):
  - Hospital Necker Enfants Malades, Paris
  - Robert Debre Hospital, Paris
  - CHU Bicetre APHP Paris Saclay, Paris
- Italy (2):
  - Aziendal Ospedaliero Universitaria Pisana Presidio Ospedale di Cisanello, Pisa, PI
  - Ospedale Bambino Gesu, Roma
- University Clinical Center Ljubljana, Ljubljana, Slovenia
- United Kingdom (2):
  - Alder Hey Childrens NHS Foundation Trust, Liverpool
  - The Royal London Childrens Hospital, London

IPD SHARING:
Plan to Share IPD: Yes